CLINICAL TRIAL: NCT04619758
Title: Emollient Therapy In Preterm & Low Birth Weight Neonates: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Abdul Ahad Jamshaid (Other)
Responsible Party: Sponsor-Investigator, Dr. Abdul Ahad Jamshaid, Senior Registrar, King Edward Medical University
Organization: King Edward Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 819/RC/KEMU
Record Dates: First submitted 2020-10-26; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Weight Gain
Keywords: Emollient Low birth weight Preterm Weight Length.
MeSH Terms: conditions — Weight Gain | interventions — Emollients; Sunflower Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emollient Group (Experimental): Mothers of the neonates in group A will be advised massage with sunflower oil.
  Interventions: Other: Emollient (sunflower oil)
- Non-Emollient Group (No Intervention): Mothers of the neonates in group B will be advised massage without any emollient.

INTERVENTIONS:
Other: Emollient (sunflower oil) — In group A, mothers will be advised to massage their babies with sunflower oil at a dose of 10 mL/kg/day twice a day in equally divided amounts. They will be called for follow up after six months of application of sunflower oil.
  Arms: Emollient Group

SUMMARY:
The objective of this study is to assess the impact of emollient therapy on gain in weight and length among preterm and low birth weight babies.

DETAILED DESCRIPTION:
The study will be conducted at the Department of Pediatric Medicine unit 1, KEMU / Mayo Hospital Lahore. Total of 140 neonates fulfilling the eligibility criteria will be enrolled. They will be randomly divided into two groups - A and B. Mothers of the neonates in group A will be advised massage with sunflower oil while mothers of the neonates in group B will be advised massage without any emollient. Babies will closely be followed up and their weight and length will be measured at six months of age and will be analyzed using SPSS v 23.0.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of both genders
* Both breast fed and non-breast fed infants
* Neonates with birth weight between 1.5 and 2.5 kg
* Preterm neonates born between 28 and 37 completed weeks of gestation

Exclusion Criteria:

* Neonates with genetic syndrome, infection or with a history of admission in NICU due to any reason will be excluded.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Six Months
  Neonates will be called for follow up after 6 months of application of sunflower oil and their weights will be measured in kilograms using digital weighing scale.
Change in Length | Six Months
  Neonates will be called for follow up after 6 months of application of sunflower oil and their lengths will be measured in centimeters using infant length scale.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul Ahad Jamshaid, FCPS MRCPCH, Principal Investigator — King Edward Medical University, Lahore, Pakistan.
Locations (1):
- King Edward Medical University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Salam RA, Darmstadt GL, Bhutta ZA. Effect of emollient therapy on clinical outcomes in preterm neonates in Pakistan: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F210-5. doi: 10.1136/archdischild-2014-307157. Epub 2015 Jan 30. PMID 25637007
- [Background] Jabraeile M, Rasooly AS, Farshi MR, Malakouti J. Effect of olive oil massage on weight gain in preterm infants: A randomized controlled clinical trial. Niger Med J. 2016 May-Jun;57(3):160-3. doi: 10.4103/0300-1652.184060. PMID 27397955
- [Background] Akhavan Karbasi S, Golestan M, Fallah R, Golshan M, Dehghan Z. Effect of body massage on increase of low birth weight neonates growth parameters: A randomized clinical trial. Iran J Reprod Med. 2013 Jul;11(7):583-8. PMID 24639794
- [Background] Kumar J, Upadhyay A, Dwivedi AK, Gothwal S, Jaiswal V, Aggarwal S. Effect of oil massage on growth in preterm neonates less than 1800 g: a randomized control trial. Indian J Pediatr. 2013 Jun;80(6):465-9. doi: 10.1007/s12098-012-0869-7. Epub 2012 Oct 4. PMID 23054851
- [Background] Salam RA, Das JK, Darmstadt GL, Bhutta ZA. Emollient therapy for preterm newborn infants--evidence from the developing world. BMC Public Health. 2013;13 Suppl 3(Suppl 3):S31. doi: 10.1186/1471-2458-13-S3-S31. Epub 2013 Dec 20. PMID 24564550